CLINICAL TRIAL: NCT02236689
Title: A Randomized, Double-blind Controlled Trial Comparing Arthroscopic Tennis Elbow Release With Arthroscopic Debridement for the Management of Chronic Lateral Epicondylitis
Brief Title: Comparing Arthroscopic Tennis Elbow Release With Arthroscopic Debridement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140553-01H
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic tennis elbow release (Active Comparator): This group will have arthroscopic tennis elbow release through a standard, two-portal technique,
  Interventions: Procedure: Arthroscopic tennis elbow release
- Non Operative (Placebo Comparator): control group will not undergo a second portal or muscle release.
  Interventions: Procedure: Non operative

INTERVENTIONS:
Procedure: Non operative — no surgical intervention
  Arms: Non Operative
Procedure: Arthroscopic tennis elbow release — Patients randomized to Arthroscopic tennis elbow release (ATER) will receive arthroscopic release of the origin of the extensor carpi radialis brevis tendon through a standard, two-portal arthroscopic technique (medial and lateral).
  Arms: Arthroscopic tennis elbow release

SUMMARY:
We propose a randomized, double-blind controlled trial comparing arthroscopic release with arthroscopic debridement for the management of chronic tennis elbow in an effort to definitively determine whether arthroscopic tennis elbow release is an effective treatment of tennis elbow, and to further provide better recommendations for the use of this procedure, in an effort to improve patient care.

DETAILED DESCRIPTION:
Lateral epicondylitis (tennis elbow) is a common occurrence in the general population with an incidence of 4-7/1000/year. More recent literature describes a 1-3% rate over the course of a lifetime, most typically affecting individuals between the ages of 35 and 50.

Tennis elbow is a common occurrence in the general population that causes lateral elbow pain and diminished grip strength, which may be debilitating. Most affected individuals achieve symptom resolution within 6 months to 1 year with measures such as physiotherapy, anti-inflammatories and corticosteroid injections, but a small subset will go on to develop chronic symptoms. Chronic tennis elbow can be treated surgically, by arthroscopic tennis elbow release (ATER), which has gained popularity in recent years as it presents a less invasive option, allows for direct visualization of the elbow joint for other pathology and has a faster return-to-work time compared to other surgical procedures. Despite its promise there have been no high quality studies evaluating the efficacy of arthroscopic tennis elbow release, bringing the actual efficacy of this procedure into question. A randomized controlled trial on arthroscopic tennis elbow release would provide much needed evidence in order to define its role in the management of tennis elbow and to help refine treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms consistent with lateral epicondylitis persisting for >6 months, and have failed conservative management
* Adult, skeletally mature (>18yrs)
* Provision of informed consent

Exclusion Criteria:

* Alternative diagnosis that better explain their symptoms
* Previous elbow trauma or surgery
* Case involving workplace insurance claims (e.g. WSIB)
* Unwilling, or unlikely in the opinion of the investigator to be followed for the duration of the study (e.g., patient refusal, unfixed address, plans to move...etc.)
* Cognitive difficulties that prevent ability to provide informed consent and reliable completion of questionnaires
* Bilateral lateral epicondylitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Mayo Elbow Performance Score | From baseline to up until 24-Months Post-Operative
  The Mayo Elbow Performance score is an outcome measure specific to the elbow to assess activities of daily living (ADLs). This outcome measure consists of 4 subscales: pain, range of motion, stability and daily function. Each section is combined for a total score out of 100 points. A higher score, indicates a better outcome.

SECONDARY OUTCOMES:
Change in Disabilities of the Arm, Shoulder and Hand (DASH) | From baseline to up until 24-Months Post-Operative
  The Disabilities of the Arm, Shoulder and Hand (DASH), is a questionnaire that measures physical function and symptoms in those with an upper extremity disorder. The DASH is a 30 item questionnaire, each question is rated using a Likert scale. The question points are combined for a total of 100 points. A higher score indicates a worse outcome.
Change in American Shoulder and Elbow Surgeons Elbow (ASES) | From baseline to up until 24-Months Post-Operative
  The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
Change in Oxford Elbow Score (OES) | From time of enrollment up until 2-years post-operative
  The Oxford Elbow Score (OES) is an outcome measure specific to patients who have had elbow surgery. The OES consists of 12 questions, looking into 3 domains: elbow function, pain, and social-psychological, using a Likert scale. Questions are summed, for a total score of 100 points. A higher score indicates a better outcome.
Change in Grip Strength | From time of enrollment up until 2-years post-operative
  Grip strength will be measured using a hand-held dynamometer. Each participant will be asked to squeeze as much as they are comfortably able for approximately 3 seconds. 3 trials will be completed on each hand. Results will be averaged, and recorded in kilograms. Higher strength is a better outcome.
Adverse Events | Ongoing from time of enrollment, up until 24-months post-operative
  Rates of study adverse events or serious adverse events (e.g. number of reoperations) will be monitored and recorded and compared between study groups. A higher rate of adverse events indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: J W Pollock, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matache BA, Berdusco R, Momoli F, Lapner PL, Pollock JW. A randomized, double-blind sham-controlled trial on the efficacy of arthroscopic tennis elbow release for the management of chronic lateral epicondylitis. BMC Musculoskelet Disord. 2016 Jun 1;17:239. doi: 10.1186/s12891-016-1093-9. PMID 27245219